CLINICAL TRIAL: NCT07002606
Title: Monitoring, Assessment, and Prevention of Potential Medication Errors in the Tertiary Healthcare Facility of Nepal: A Mixed-method Study
Brief Title: The General Objective of This Study is to Monitor, Assess, and Prevent the Potential Medication Errors Among Inpatients in the Tertiary Healthcare Facility of Nepal. This Study Aims to Develop and Implement the Medication Errors Reporting System in Hospital Settings.
Status: Not yet recruiting | Type: Observational
Sponsor: Kathmandu University School of Medical Sciences (Other)
Responsible Party: Principal Investigator, Rudip Thapa, Assistant Professor (Pharmacology), Kathmandu University School of Medical Sciences
Other Study IDs: 147/24; PhD- 80/8 t-HS-04 (Other Grant/Funding Number: University Grant Commission)
Record Dates: First submitted 2025-05-25; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Prescription With Medication Errors
Keywords: Medication errors; Mixed method study; tertiary healthcare facility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: medication errors reporting guidelines — the intervention is designed to reduce the medication errors and develop the culture of reporting the Medication errors in clinical settings.

SUMMARY:
The goal of this observational study is to develop and implement Medication errors reporting system using the error reporting guidelines. The main question it aims to answer is:

"Does development and implementation of Medication errors reporting guideline will help to reduce the errors rate and improve the patient safety?"

ELIGIBILITY:
Inclusion Criteria:

* For the quantitative part, the inclusion criteria are patients of all age groups and prescriptions issued to inpatients.
* For the qualitative part of the study, inclusion criteria are healthcare professionals aged more than 18 years working in Dhulikhel Hospital.

Exclusion criteria:

* The exclusion criteria will be incomplete and unclear prescriptions.
* The healthcare persons who accepted the consent but couldn't complete the survey will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Healthcare professionals including Doctors, Nurses and Pharmacist who are working in Dhulikhel Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
reduction in Mediation error rate | 6 months after the implementation of the Medication errors reporting guidelines
  The newly developed Medication errors reporting guidelines will be implemented and will be used to evaluate the reduction in medication errors incident rates.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sony Shakya Professor in Pharmacology, PhD, Study Director — Kathmandu University School of Medical Science

IPD SHARING:
Plan to Share IPD: No